CLINICAL TRIAL: NCT04375397
Title: IbrutiNib in SARS CoV-2 Induced Pulmonary Injury and Respiratory Failure (iNSPIRE)
Brief Title: Study of Oral Ibrutinib Capsules to Assess Respiratory Failure in Adult Participants With Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) and Pulmonary Injury
Acronym: iNSPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Janssen Research & Development LLC; Pharmacyclics LLC (An AbbVie Company) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M20-310
Record Dates: First submitted 2020-05-04; First posted 2020-05-05 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: CoronaVirus Induced Disease-2019 (COVID-19)
Keywords: CoronaVirus Induced Disease-2019; COVID-19; Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2); Pulmonary Injury; Ibrutinib; Imbruvica; Respiratory failure
MeSH Terms: conditions — COVID-19; Lung Injury; Respiratory Insufficiency | interventions — ibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ibrutinib 420 mg + SOC (Experimental): 420 mg ibrutinib administered once daily as three hard gelatin capsules (140 mg each) with approximately 240 mL of water for up to 28 days and supportive care (standard-of-care, SOC)
  Interventions: Drug: Ibrutinib
- Placebo + SOC (Placebo Comparator): Three hard gelatin placebo capsules administered once daily with approximately 240 mL of water for up to 28 days and supportive care (standard-of-care, SOC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibrutinib — Capsules were to be administered orally with water once daily. For participants who required nasogastric tube (NGT) placement while on study, capsules may have been administered by opening the capsules, mixing with water, and flushing down the NGT.
  Other Names: Imbruvica
  Arms: Ibrutinib 420 mg + SOC
Drug: Placebo — Capsules were to be administered orally with water once daily. For participants who required nasogastric tube (NGT) placement while on study, capsules may have been administered by opening the capsules, mixing with water, and flushing down the NGT.
  Arms: Placebo + SOC

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Lung failure is the main cause of death related to COVID-19 infection. The main objective of this study was to evaluate if ibrutinib is safe and can reduce respiratory failure in participants with COVID-19 infection.

DETAILED DESCRIPTION:
This was a Phase 2, multicenter, randomized, placebo-controlled, double-blind study to evaluate the addition of ibrutinib to supportive care in hospitalized participants who presented with COVID-19- related pulmonary distress requiring supplemental oxygen. Participants were randomized in a 1:1 ratio to receive placebo + supportive care, denoted as SOC or standard-of-care, or ibrutinib 420 mg + SOC, with randomization stratified by prescription for remdesivir.

Participants were to be treated with either placebo or ibrutinib in addition to supportive care for up to 28 days unless they met treatment discontinuation criteria and were to be followed for 58 days following start of therapy or until death, whichever occurred first. Treatment could have been stopped at the discretion of the treating physician after 14 days if the participant was clinically stable and had been off supplemental oxygen for > 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Requires hospitalization for COVID-19 infection
* Has Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by reverse transcription polymerase chain reaction (RT-PCR) test before study entry
* Requires supplemental oxygen for pulmonary distress related to COVID-19 infection, and has been on supplemental oxygen for no more than 5 days, and on breathing room air have oxygen saturation levels of 94% or less
* Has radiographic evidence of pulmonary infiltrates
* Females of childbearing potential (FCBP) must use 1 reliable form of contraception or have complete abstinence from heterosexual intercourse during the following time periods related to this study: while participating in the study; and for at least 1 month after discontinuation of study drug. FCBP must be referred to a qualified provider of contraceptive methods if needed. FCBP must have a negative serum pregnancy test as of screening.
* Men must agree to use a latex condom during treatment and for up to 3 months after the last dose of ibrutinib during sexual contact with a FCBP.
* Adequate hematologic, hepatic and renal function as described in the protocol
* Must be within 10 days of confirmed diagnosis of COVID-19

Exclusion Criteria:

* Respiratory failure at time of screening as defined per protocol with any of these following therapies:

  * Endotracheal intubation and mechanical ventilation
  * Extracorporeal membrane oxygenation (ECMO)
  * High flow nasal cannula oxygen at flow rates ≥ 30 L/min and fraction of delivered oxygen ≥ 0.5
  * Non-invasive positive pressure ventilation
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* On a Bruton's tyrosine kinase (BTK)-inhibitor, anti-interleukin 6 (IL6), anti-interleukin 6R (IL6R), or Janus kinase inhibitor (JAKi)
* Has received rituximab within 180 days from study entry.
* Known bleeding disorders
* Major surgery within 4 weeks of study entry
* Participants in whom surgery is anticipated to be necessary within 72 hours
* History of stroke or bleeding around or within brain within 6 months prior to enrollment
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV)
* Currently active, clinically significant cardiovascular disease
* Asymptomatic arrythmias and or history of ejection fraction < 40% on an echo
* Participants receiving a strong cytochrome P450 (CYP) 3A4 inhibitor with the exception of those receiving anti-fungal therapy/prophylaxis
* Chronic liver disease and hepatic impairment meeting Child Pugh class C
* Female participants who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or within 1 month of last dose of study drug. Male participants who plan to father a child while enrolled in this study or within 3 months after the last dose of study drug.
* Unwilling or unable to participate in all required study evaluations and procedures
* Vaccinated with a live, attenuated vaccine within 4 weeks
* Uncontrolled high blood pressure
* On therapeutic anticoagulation at baseline
* Participants with cancer, history of interstitial lung disease, and/or history of malignancies as defined in the protocol
* Co-enrolled in another interventional trial
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3.0 × ULN, and total bilirubin > 2.0 × ULN
* International normalized ratio (INR) ≥ 1.5 × ULN attributable to coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (9):
- United States (9):
  - Stanford University School of Med /ID# 221954, Stanford, California
  - Medstar Washington Hospital Center /ID# 221886, Washington D.C., District of Columbia
  - Duplicate_GW Medical Faculty Associates /ID# 222023, Washington D.C., District of Columbia
  - Midway Immunology and Research /ID# 222004, Ft. Pierce, Florida
  - University of Miami /ID# 223227, Miami, Florida
  - Triple O Research Institute /ID# 222944, West Palm Beach, Florida
  - Brigham & Women's Hospital /ID# 221847, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 222994, Boston, Massachusetts
  - Intermountain Healthcare /ID# 221955, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Requests for access to individual participant data from ibrutinib clinical studies conducted by AbbVie can be submitted through Yale Open Data Access (YODA) Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu/

REFERENCES:
- [Derived] Coutre SE, Barnett C, Osiyemi O, Hoda D, Ramgopal M, Fort AC, Qaqish R, Hu Y, Ninomoto J, Alami NN, Styles L, Treon SP. Ibrutinib for Hospitalized Adults With Severe Coronavirus Disease 2019 Infection: Results of the Randomized, Double-Blind, Placebo-Controlled iNSPIRE Study. Open Forum Infect Dis. 2022 Mar 24;9(5):ofac104. doi: 10.1093/ofid/ofac104. eCollection 2022 May. PMID 35493119

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Period: Overall Study
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Started | 22 | 24
Completed | 13 | 18
Not Completed | 9 | 6
Not completed — Death | 1 | 1
Not completed — Withdrew consent | 2 | 0
Not completed — Lost to Follow-up | 6 | 4
Not completed — Other, not specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.52) | 55.2 (11.73) | 52.8 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 12 | 26
  Black or African American | 4 | 4 | 8
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Multiple | 0 | 0 | 0
  Other | 0 | 0 | 0
  Missing | 4 | 6 | 10
COVID-19 symptom onset duration prior to baseline (days) [Mean (Standard Deviation); unit: days] — Baseline refers to the last non-missing observation on or before the first day of study drug administration.
  days | 9.27 (2.567) | 9.08 (2.765) | 9.17 (2.644)
Number of participants with a score of 4 on the WHO-8 ordinal scale at screening [Count of Participants; unit: Participants] — WHO-8 scores: 0 (uninfected); 1 (ambulatory, no limitation of activities); 2 (ambulatory, limitation of activities); 3 (hospitalized with mild disease, no oxygen therapy); 4 (hospitalized with mild disease, oxygen by mask or nasal prongs); 5 (hospitalized with severe disease, non-invasive ventilation or high-flow oxygen); 6 (hospitalized with severe disease, intubation and mechanical ventilation); 7 (hospitalized with severe disease, ventilation and additional organ support [pressors, renal replacement therapy, extracorporeal membrane oxygenation]); and 8 (death).
  Participants | 22 | 24 | 46
Stratification factor of prescription for remdesivir [Count of Participants; unit: Participants]
  Yes | 13 | 16 | 29
  No | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive and Without Respiratory Failure Through Day 28
Description: Respiratory failure is defined as a clinical diagnosis of respiratory failure and initiation of one of the following therapies: endotracheal intubation and mechanical ventilation; OR extracorporeal membrane oxygenation; OR high-flow nasal cannula oxygen delivery (i.e., reinforced nasal cannula delivering heated, humidified oxygen with fraction of delivered oxygen ≥ 0.5 and flow rates of ≥ 30 L/min); OR non-invasive positive pressure ventilation; OR clinical diagnosis of respiratory failure with initiation of none of these measures only when clinical decision-making is driven solely by resource limitation.
Time Frame: Through Day 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
percentage of participants | 86.4 [74.4 to 93.2] | 79.2 [66.9 to 87.7]
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; The difference in response rates between the experimental arm and the control arm were analyzed using the Miettinen-Nurminen (MN) method, adjusting for the stratification factor of prescription for remdesivir. The MN test p-value for testing the rate difference = 0 at two-sided alpha = 0.2; Test type: Superiority; p = 0.599, Miettinen-Nurminen method; Adjusted risk difference (%) = 5.8, 80% CI 2-sided [-9.2 to 20.4] — Ibrutinib 420 mg + SOC - Placebo + SOC Miettinen-Nurminen (MN) CI for the adjusted risk difference across strata
Statistical Analysis 2: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; The difference in response rates between the experimental arm and the control arm were analyzed using the Miettinen-Nurminen (MN) method, adjusting for the stratification factor of prescription for remdesivir. The MN test p-value for testing the rate difference = 0 at twosided alpha = 0.2; Test type: Superiority; p = 0.599, Miettinen-Nurminen method; Adjusted risk difference (%) = 5.8, 95% CI 2-sided [-18.1 to 28.7] — Ibrutinib 420 mg + SOC - Placebo + SOC Miettinen-Nurminen (MN) CI for the adjusted risk difference across strata

2. Secondary Outcome: Change in the World Health Organization (WHO)-8 Ordinal Scale From Baseline at Study Day 14
Description: The WHO-8 is an ordinal scale for clinical improvement with scores ranging from 0 to 8, where a lower score indicates better clinical status. A score of 0 represents uninfected; 1 (ambulatory, no limitation of activities); 2 (ambulatory, limitation of activities); 3 (hospitalized with mild disease, no oxygen therapy); 4 (hospitalized with mild disease, oxygen by mask or nasal prongs); 5 (hospitalized with severe disease, non-invasive ventilation or high-flow oxygen); 6 (hospitalized with severe disease, intubation and mechanical ventilation); 7 (hospitalized with severe disease, ventilation and additional organ support [pressors, renal replacement therapy, extracorporeal membrane oxygenation]); and 8 (death). Negative values indicate improvement from baseline.
Time Frame: At Day 14
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug; participants with baseline and Day 14 score data
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
Participants
  -4 points | 2 | 3
  -3 points | 12 | 9
  -2 points | 5 | 7
  -1 point | 0 | 2
  0 points | 1 | 1
  1 point | 1 | 1
  3 points | 1 | 1
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Change in ordinal score from baseline to day 14 = -3 To evaluate the odds of clinical status improvement as determined by the WHO-8 ordinal scale, a multinomial logistic regression model was used. Pairwise Comparison in Reference to the Group with Change = -4; Test type: Superiority; p = 0.886, Multinomial Logistic Regression; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.13 to 10.44]
Statistical Analysis 2: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Change in ordinal score from baseline to day 14 = -2 To evaluate the odds of clinical status improvement as determined by the WHO-8 ordinal scale, a multinomial logistic regression model was used. Pairwise Comparison in Reference to the Group with Change = -4; Test type: Superiority; p = 0.705, Multinomial Logistic Regression; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.06 to 6.43]
Statistical Analysis 3: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Change in ordinal score from baseline to day 14 = -1 To evaluate the odds of clinical status improvement as determined by the WHO-8 ordinal scale, a multinomial logistic regression model was used. Pairwise Comparison in Reference to the Group with Change = -4; Test type: Superiority; p = 0.996, Multinomial Logistic Regression; Odds Ratio (OR) = 0.00, 95% CI 2-sided [lower limit 0.00] (The upper limit of this 95% CI is infinite.)
Statistical Analysis 4: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Change in ordinal score from baseline to day 14 = 0 To evaluate the odds of clinical status improvement as determined by the WHO-8 ordinal scale, a multinomial logistic regression model was used. Pairwise Comparison in Reference to the Group with Change = -4; Test type: Superiority; p = 0.969, Multinomial Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.04 to 32.18]
Statistical Analysis 5: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Change in ordinal score from baseline to day 14 = 1 To evaluate the odds of clinical status improvement as determined by the WHO-8 ordinal scale, a multinomial logistic regression model was used. Pairwise Comparison in Reference to the Group with Change = -4; Test type: Superiority; p = 0.969, Multinomial Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.04 to 32.18]
Statistical Analysis 6: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Change in ordinal score from baseline to day 14 = 3 To evaluate the odds of clinical status improvement as determined by the WHO-8 ordinal scale, a multinomial logistic regression model was used. Pairwise Comparison in Reference to the Group with Change = -4; Test type: Superiority; p = 0.969, Multinomial Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.04 to 32.18]

3. Secondary Outcome: Median Reduction in Days Spent on Supplemental Oxygen
Description: Days spent on supplemental oxygen was set as the date of the participant being off of supplemental oxygen minus the date of initiation of supplemental oxygen + 1 day. If a participant received more than 1 period of supplemental oxygen therapy during the study or switched from supplemental oxygen to a more intensive therapy, then the days spent on supplemental oxygen were to be calculated as the sum of all the periods where the participant was on supplemental oxygen or a more intensive therapy through Day 28. If the date of the first initiation of supplemental oxygen was before Baseline Day 1, then the days spent on supplemental oxygen were to be calculated from Baseline Day 1 to the date of the participant being off the supplemental oxygen. Time on supplemental oxygen was to be imputed to the maximum number of days on study drug (28) for all points following the death of a participant.
Time Frame: Up to Day 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Measure: Median (Full Range); unit: days
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
days | 5.0 [1 to 28] | 6.5 [1 to 21]
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Median days spent on supplemental oxygen was compared between treatment groups using Van Elteren's test with the stratification factor of prescription for remdesivir; Test type: Superiority; p = 0.801, Van Elteren's test; Difference in Medians = -1.5 — Ibrutinib 420 mg + SOC - Placebo + SOC

4. Secondary Outcome: All-Cause Mortality at Study Days 7, 14, 21, and 28
Description: The percentage of participants with mortality from any cause was recorded.
Time Frame: At Study Days 7, 14, 21, and 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
percentage of participants
  Day 7 | 0 [0.0 to 6.9] | 0 [0.0 to 6.4]
  Day 14 | 0 [0.0 to 6.9] | 0 [0.0 to 6.4]
  Day 21 | 4.5 [1.4 to 14.0] | 0 [0.0 to 6.4]
  Day 28 | 4.5 [1.4 to 14.0] | 0 [0.0 to 6.4]
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; At Day 7-- Ibrutinib 420 mg + SOC - Placebo + SOC The Miettinen-Nurminen (MN) test p-value for testing the rate difference = 0 adjusting for the stratification factor of prescription for remdesivir using Cochran-Mantel-Haenszel weights at two-sided alpha of 0.2 and associated confidence intervals are reported; Test type: Superiority; p = 1.000, Miettinen-Nurminen; Mortality rate difference = 0.0, 80% CI 2-sided [-6.7 to 7.3]
Statistical Analysis 2: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 1.000, Miettinen-Nurminen; Mortality rate difference = 0.0, 95% CI 2-sided [-14.4 to 15.5]
Statistical Analysis 3: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; At Day 14-- Ibrutinib 420 mg + SOC - Placebo + SOC The Miettinen-Nurminen (MN) test p-value for testing the rate difference = 0 adjusting for the stratification factor of prescription for remdesivir using Cochran-Mantel-Haenszel weights at two-sided alpha of 0.2 and associated confidence intervals are reported; Test type: Superiority; p = 1.000, Miettinen-Nurminen; Mortality rate difference = 0.0, 80% CI 2-sided [-6.7 to 7.3]
Statistical Analysis 4: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 1.000, Miettinen-Nurminen; Mortality rate difference = 0.0, 95% CI 2-sided [-14.4 to 15.5]
Statistical Analysis 5: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; At Day 21-- Ibrutinib 420 mg + SOC - Placebo + SOC The Miettinen-Nurminen (MN) test p-value for testing the rate difference = 0 adjusting for the stratification factor of prescription for remdesivir using Cochran-Mantel-Haenszel weights at two-sided alpha of 0.2 and associated confidence intervals are reported; Test type: Superiority; p = 0.267, Miettinen-Nurminen; Mortality rate difference = 4.8, 80% CI 2-sided [-1.7 to 14.8]
Statistical Analysis 6: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.267, Miettinen-Nurminen; Mortality rate difference = 4.8, 95% CI 2-sided [-9.6 to 22.8]
Statistical Analysis 7: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; At Day 28-- Ibrutinib 420 mg + SOC - Placebo + SOC The Miettinen-Nurminen (MN) test p-value for testing the rate difference = 0 adjusting for the stratification factor of prescription for remdesivir using Cochran-Mantel-Haenszel weights at two-sided alpha of 0.2 and associated confidence intervals are reported; Test type: Superiority; p = 0.267, Miettinen-Nurminen; Mortality rate difference = 4.8, 80% CI 2-sided [-1.7 to 14.8]
Statistical Analysis 8: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; [analysis description as in outcome 4, analysis 7]; Test type: Superiority; p = 0.267, Miettinen-Nurminen; Mortality rate difference = 4.8, 95% CI 2-sided [-9.6 to 22.8]

5. Secondary Outcome: Percentage of Participants Experiencing Respiratory Failure or Death on Study Days 7, 14, 21, and 28
Description: Respiratory failure is defined as a clinical diagnosis of respiratory failure and initiation of one of the following therapies: endotracheal intubation and mechanical ventilation; OR extracorporeal membrane oxygenation; OR high-flow nasal cannula oxygen delivery (i.e., reinforced nasal cannula delivering heated, humidified oxygen with fraction of delivered oxygen ≥ 0.5 and flow rates of ≥ 30 L/min), OR non-invasive positive pressure ventilation; OR clinical diagnosis of respiratory failure with initiation of none of these measures only when clinical decision-making is driven solely by resource limitation.
Time Frame: At Study Days 7, 14, 21, and 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
percentage of participants
  Day 7 | 9.1 [3.8 to 20.0] | 20.8 [12.3 to 33.1]
  Day 14 | 9.1 [3.8 to 20.0] | 20.8 [12.3 to 33.1]
  Day 21 | 13.6 [6.8 to 25.6] | 20.8 [12.3 to 33.1]
  Day 28 | 13.6 [6.8 to 25.6] | 20.8 [12.3 to 33.1]
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Failure/Mortality Rate Difference Compared to Placebo + SOC at Day 7 The difference in response rates between the experimental arm and the control arm was analyzed using the Miettinen-Nurminen (MN) method adjusting for the stratification factor of prescription for remdesivir. MN test p-value for testing the rate difference = 0 adjusting for the stratification factor of prescription for remdesivir using Cochran-Mantel-Haenszel weights at two-sided alpha of 0.2; Test type: Superiority; p = 0.314, Miettinen-Nurminen; Adjusted risk difference (%) = -10.7, 80% CI 2-sided [-24.8 to 3.3]
Statistical Analysis 2: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.314, Miettinen-Nurminen; Adjusted risk difference (%) = -10.7, 95% CI 2-sided [-32.8 to 12.0]
Statistical Analysis 3: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Failure/Mortality Rate Difference Compared to Placebo + SOC at Day 14 The difference in response rates between the experimental arm and the control arm was analyzed using the Miettinen-Nurminen (MN) method adjusting for the stratification factor of prescription for remdesivir. MN test p-value for testing the rate difference = 0 adjusting for the stratification factor of prescription for remdesivir using Cochran-Mantel-Haenszel weights at two-sided alpha of 0.2; Test type: Superiority; p = 0.314, Miettinen-Nurminen; Adjusted risk difference (%) = -10.7, 80% CI 2-sided [-24.8 to 3.3]
Statistical Analysis 4: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.314, Miettinen-Nurminen; Adjusted risk difference (%) = -10.7, 95% CI 2-sided [-32.8 to 12.0]
Statistical Analysis 5: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Failure/Mortality Rate Difference Compared to Placebo + SOC at Day 21 The difference in response rates between the experimental arm and the control arm was analyzed using the Miettinen-Nurminen (MN) method adjusting for the stratification factor of prescription for remdesivir. MN test p-value for testing the rate difference = 0 adjusting for the stratification factor of prescription for remdesivir using Cochran-Mantel-Haenszel weights at two-sided alpha of 0.2; Test type: Superiority; p = 0.599, Miettinen-Nurminen; Adjusted risk difference (%) = -5.8, 80% CI 2-sided [-20.4 to 9.2]
Statistical Analysis 6: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.599, Miettinen-Nurminen; Adjusted risk difference (%) = -5.8, 95% CI 2-sided [-28.7 to 18.1]
Statistical Analysis 7: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Failure/Mortality Rate Difference Compared to Placebo + SOC at Day 28 The difference in response rates between the experimental arm and the control arm was analyzed using the Miettinen-Nurminen (MN) method adjusting for the stratification factor of prescription for remdesivir. MN test p-value for testing the rate difference = 0 adjusting for the stratification factor of prescription for remdesivir using Cochran-Mantel-Haenszel weights at two-sided alpha of 0.2; Test type: Superiority; p = 0.599, Miettinen-Nurminen; Adjusted risk difference (%) = -5.8, 80% CI 2-sided [-20.4 to 9.2]
Statistical Analysis 8: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.599, Miettinen-Nurminen; Adjusted risk difference (%) = -5.8, 95% CI 2-sided [-28.7 to 18.1]

6. Secondary Outcome: Mechanical Ventilation-Free Survival
Description: Mechanical ventilation-free survival is defined as the number of days from Baseline Day 1 to the date when a participant initiated mechanical ventilation or died, whichever occurred first, during the 28 days post baseline. If the specified event did not occur by Day 28, participants were to be censored. Specifically, a participant without any post-baseline assessment record was to be censored at Baseline Day 1, a participant who prematurely discontinued from study without a record of death or start of mechanical ventilation was to be censored at the earlier timepoint of the date of study discontinuation or Day 28, an ongoing participant in the study without a record of death or start of mechanical ventilation was to be censored at the earlier timepoint of the date of the last evidence that the participant is not on mechanical ventilation or Day 28.
Time Frame: Up to Day 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
days | NA [NA to NA] — Not calculable/estimable due to low number of participants with events | NA [NA to NA] — Not calculable/estimable due to low number of participants with events
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; For the analysis of mechanical ventilation-free survival, the distribution of time to event was estimated by treatment group using Kaplan-Meier methodology and compared between the experimental arm and the control arm using the log-rank test stratified by prescription for remdesivir; Test type: Superiority; p = 0.851, Log Rank

7. Secondary Outcome: Days on Mechanical Ventilation
Description: Days spent on mechanical ventilation was defined as the date of the participant being off mechanical ventilation - date of initiation of mechanical ventilation + 1 day. If a participant received more than 1 period of mechanical ventilation during the study or switched from mechanical ventilation to a more intensive therapy, then the days spent on mechanical ventilation were to be calculated as the sum of all the periods where the participant is on mechanical ventilation or a more intensive therapy through Day 28.
Time Frame: Up to Day 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Measure: Median (Full Range); unit: days
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
days | 0.0 [0 to 28] | 0.0 [0 to 28]
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Median days spent on mechanical ventilation were compared between treatment groups using Van Elteren's test with the stratification factor of prescription for remdesivir; Test type: Superiority; p = 0.745, Van Elteren's test; Difference in Medians = 0.0 — Ibrutinib 420 mg + SOC - Placebo + SOC

8. Secondary Outcome: Median Duration of Hospitalization
Description: Median duration of hospitalization is defined as the hospitalization discharge date - hospitalization admission date + 1 day. If a participant was hospitalized more than once during the study then the hospitalization time was to be calculated as the sum of all the periods when the participant was hospitalized through Day 28.
Time Frame: Up to Day 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Measure: Median (Full Range); unit: days
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
days | 6.0 [2 to 28] | 6.5 [3 to 28]
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; Median duration of hospitalization was compared between treatment groups using Van Elteren's test with the stratification factor of prescription for remdesivir; Test type: Superiority; p = 0.977, Van Elteren's test]; Difference in Medians = -0.5 — Ibrutinib 420 mg + SOC - Placebo + SOC

9. Secondary Outcome: Time to Discharge From Hospital
Description: Time to discharge from hospital is defined as the number of days from Baseline Day 1 to the date of the last evidence that a participant is last discharged from hospital, during the 28 days post baseline. If the specified event did not occur by Day 28, participants were censored. Specifically, a participant without any postbaseline assessment record was to be censored at Baseline Day 1, a participant who died was to have time to discharge from hospital censored at Day 28, a participant who prematurely discontinued from study without a record of hospitalization discharge was to be censored at the earlier timepoint of the date of study discontinuation or Day 28, an on-going participant in the study without a record of hospitalization discharge was to be censored at the earlier timepoint of the date of the last evidence that the participant is hospitalized or Day 28.
Time Frame: Up to Day 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug
Measure: Median (Full Range); unit: days
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
days | 6.0 [5.0 to 10.0] | 6.5 [5.0 to 9.0]
Statistical Analysis 1: Comparison: Ibrutinib 420 mg + SOC vs Placebo + SOC; For the analysis of time to discharge from hospital, the distribution of time to event was estimated by treatment group using Kaplan-Meier methodology and compared between the experimental arm and the control arm using the log-rank test stratified by prescription for remdesivir; Test type: Superiority; p = 0.969, Log Rank

10. Secondary Outcome: Partial Pressure of Oxygen in Arterial Blood (PaO2) to Fraction of Inspired Oxygen (FiO2) Ratio
Description: The PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2). A PaO2/FiO2 ratio of 300 to 200 is mild, 200 to 100 moderate, and <100 is severe Adult Respiratory Distress Syndrome (ARDS).
Time Frame: At Study Days 7, 14, 21, and 28
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug. Participants with non-missing baseline and at least one post-baseline value are included in the analyses.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 2 | 3
mmHg
  Day 7 | 100 (56.07) | 87 (33.35)
  Day 14: number analyzed (Participants) | 0 | 0
  Day 21: number analyzed (Participants) | 1 | 0
  Day 21 | 269 |
  Day 28: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Oxygenation Index
Description: The oxygenation index is used to assess the intensity of ventilatory support required to maintain oxygenation. An index of 0 to < 25 is predictive of a good outcome; 25 to <40 indicates a chance of death >40%; and an index of 40 to 1000 warrants consideration of extracorporeal membrane oxygenation (ECMO).
Time Frame: At Study Days 7, 14, 21, and 28
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 2 | 2
units on a scale
  Day 7: number analyzed (Participants) | 1 | 0
  Day 7 | 14 |
  Day 14: number analyzed (Participants) | 1 | 1
  Day 14 | 19 | 12
  Day 21 | 33 (43.61) | 20 (1.75)
  Day 28: number analyzed (Participants) | 0 | 2
  Day 28 |  | 12 (4.26)

12. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events (TEAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to 70 days)
Population: Safety Population: all participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 22 | 24
Participants | 12 | 12

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to the end of study; median time on follow-up was Ibrutinib 420 mg + SOC (58.0 days); and Placebo + SOC (62.0 days). Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 30 days after last dose, up to 70 days.
Description: All-cause mortality and adverse events: all participants who received at least one dose of study drug
Arm/Group | Ibrutinib 420 mg + SOC | Placebo + SOC
All-Cause Mortality (participants affected / at risk) | 1/22 | 1/24
Serious Adverse Events (participants affected / at risk) | 4/22 | 3/24
Other Adverse Events (participants affected / at risk) | 8/22 | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib 420 mg + SOC (N=22) | Placebo + SOC (N=24)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (2)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 2 (2)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib 420 mg + SOC (N=22) | Placebo + SOC (N=24)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (2)
HYPERTENSION (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT04375397/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT04375397/SAP_001.pdf